CLINICAL TRIAL: NCT07197840
Title: Chronic Subdural Hematoma Treated With Numen SILK Coiling of Middle Meningeal Artery
Brief Title: The CHALLENGER Registry
Acronym: CHALLENGER
Status: Not yet recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shahram Majidi, Associate Professor of Neurosurgery, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-25-00525
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Subdural Hemorrhage (cSDH)
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Numen SILK: Patients treated with the Numen SILK coil embolization system
  Interventions: Device: Numen SILK coil embolization system

INTERVENTIONS:
Device: Numen SILK coil embolization system — The Numen SILK coil embolization system is designed to be used in conjunction with the NumenFR detachment system. It consists of two main parts: • Introducer Sheath: The purpose of this sheath is to facilitate the introduction of the coil into the microcatheter. • Coil System: Composed of the pusher and coil implant. The coil is a permanent implant intended to occlude blood flow in vascular abnormalities. The pusher is used to deliver the coil implant to the target lesion. The NumenFR detachment system is a sterile, handheld, single-patient use device designed for use with the Numen SILK coil embolization system and is operated by two pre-loaded batteries

SUMMARY:
The study is a multi-center prospective, single-arm, post-market study evaluating the efficacy and radiologic and functional outcomes associated use of the Numen SILK coils for Middle Meningeal Artery (MMA) embolization following Chronic Subdural Hematoma (cSDH) compared to surgical evacuation or medical management alone.

Chronic subdural hematoma is a collection of blood between the dural mater and the brain. It typically develops over time in older adults or people on anticoagulant medication. Blood slowly accumulates over time and often becomes encapsulated by a fibrous membrane over weeks or months, which can lead to the gradual development of symptoms. Middle Meningeal Artery embolization (MMAE) through coiling provides a minimally invasive option for cSDH treatment and prevention of reaccumulation and recurrence.

DETAILED DESCRIPTION:
The NumenFR detachment system is a sterile, handheld, single-patient use device designed for use with the Numen SILK coil embolization system and is operated by two pre-loaded batteries. The analysis of the Numen SILK coil embolization system will occur prospectively if it is determined the patient meets the enrollment criteria. All patients enrolled in the study will receive supportive and medical treatment by choice of the treating physician and in accordance with standard of care. Such treatment includes but is not limited to: neurointensive care, neuromonitoring, and surgical and medical management of cSDH.

ELIGIBILITY:
* Age 18-98 years inclusively
* Per CT of the head, (one of the following):

  * Unilateral convexity cSDH measuring at least 10 mm in thickness OR
  * Bilateral cSDH if only one side is considered for treatment and the contralateral side is asymptomatic and < 5 mm in thickness.
* cSDH at least 2/3 isodense or hypodense, verified on axial CT slice used to measure the thickness of the qualifying cSDH
* Qualifying baseline head CT performed within the 14 days prior to treatment
* Patient or legally authorized representative agrees to be participated in the study and provides written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Secondary cause apart from trauma for the qualifying SDH, such as an underlying vascular abnormality or tumor
* Bilateral cSDH with unknown origin of symptoms
* Participants who underwent prior embolization of either MMA
* Tentorial or interhemispheric SDH
* mRS >4
* On tranexamic acid
* Intractable coagulation dysfunction or abnormal platelet count and function (pre-operative International Normalized Ratio [INR] > 1.5 and/or platelet count < 80109/L)
* Anatomical variations that may affect the safety of MMA embolization (e.g., prominent middle MMA ophthalmic artery anastomosis)
* Known contraindications to angiography
* Known intolerance to occlusion procedures
* Known vascular anatomy (small artery size) or blood flow (high vascular resistance peripheral to the feeding arteries) that precludes catheter placement or coil embolization
* Known presence of collateral vessel pathways potentially endangering normal territories or cranial nerves during embolization.
* Known large diameter arteriovenous shunt, i.e., where the blood does not pass through an arterial/capillary/venous transition but directly from an artery to a vein or presence of patent extra-to-intracranial anastomoses (where study embolization devices could pass directly into the internal carotid artery, vertebral artery, or intracranial vasculature) that cannot be addressed with coil embolization.
* Patient has a known active systemic infection or sepsis
* Patient is pregnant, planning to become pregnant, or lactating
* Life expectancy of less than 6 months due to comorbid terminal conditions
* Concurrent participation in another research protocol for investigation of an experimental therapy
* Known or suspected to not be able to comply with the study protocol

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population for this study will be comprised of up to 100 patients with chronic subdural hematoma (cSDH).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that need rescue surgery or die within 180 days of MMA coil embolization | 180 days
  The proportion of patients centrally deemed to need rescue surgery or die within 180 days of MMA coil embolization

SECONDARY OUTCOMES:
Recurrent or residual chronic subdural hematoma measuring greater than 10 mm in thickness | 180 days
  Recurrent or residual chronic subdural hematoma at 180 days measuring greater than 10 mm in thickness
Number of patients requiring reoperation or surgical rescue within | 180 days
  Number of patients requiring reoperation or surgical rescue within 180 days
Worsening of or death from neurological causes within 180 days | 180 days
  Worsening of or death from neurological causes within 180 days
Major disabling stroke from neurological causes within 180 days | 180 days
  Major disabling stroke from neurological causes within 180 days
Rate of serious adverse events from neurological causes within 180 days | 180 days
  Rate of serious adverse events from neurological causes within 180 days
Change in hematoma thickness | Baseline, at 90 days and at 180 days
  Change in hematoma thickness from baseline to the repeat scan at 90 days and from baseline to the repeat scan at 180 days
Modified Rankin Scale (mRS) score at 90 days and at 180 days | at 90 days and at 180 days
  Modified Rankin Scale score at 6 months will be collected to determine patient functional outcomes at 6 months. The scale runs from 0-6, running from perfect health without symptoms to death:
  * 0 - No symptoms.
  * 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
  * 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * 3 - Moderate disability. Requires some help, but able to walk unassisted.
  * 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * 6 - Dead.
Number of target MMA injuries related to study device | 180 days
  The number of injuries to the target middle meningeal artery (MMA) that are determined to be related to the study device, as identified through adverse event reporting during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Majidi, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Upon the completion of the study, Mount Sinai's data management team will clean and analyze all data in preparation of manuscript writing and publication. The intention will be to publish together between the principal investigator and the sponsor. Following publication, Mount Sinai will archive and store all associated data on its cloud-based system.